CLINICAL TRIAL: NCT05136235
Title: Pulmonary Hypertension in Extremely Preterm Infants - A Prospective Cohort Study
Brief Title: Pulmonary Hypertension in Extremely Preterm Infants
Acronym: PiEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: AZ Sint-Jan AV (Other); Universitaire Ziekenhuizen KU Leuven (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Ziekenhuis Oost-Limburg (Other); University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PiEP study
Record Dates: First submitted 2021-10-06; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-10

CONDITIONS: Bronchopulmonary Dysplasia; Pulmonary Hypertension; Premature Birth
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypertension, Pulmonary; Premature Birth | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extremely preterm newborns (Other): All extremely preterm newborns in Flanders will be included, it is a single arm study
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: NT-proBNP

INTERVENTIONS:
Diagnostic Test: Echocardiography — There will be screened for pulmonary hypertension by means of serial echocardiographies during the study period
Diagnostic Test: NT-proBNP — At 36 weeks postmenstrual age there will be screened for pulmonary hypertension by means of an NT-proBNP measurement in a blood sample

SUMMARY:
Extremely preterm infants are at risk for developing bronchopulmonary dysplasia (BPD) and associated chronic pulmonary hypertension (PH), a consequence of altered pulmonary vasculature. This condition occurs in about 25% of babies with BPD, and the association grows with increasing BPD severity. Other risk factors have been described as well. Morbidity and mortality associated with prematurity and/or BPD increase significantly in the presence of PH.

Thus, international guidelines encourage the use of standardized screening protocols for this condition. However, several questions regarding these recommendations are left unanswered, such as a clear definition for PH in this population.

The research aim is to prospectively evaluate prevalence, risk factors and clinical course of PH in these children. The investigators aim to identify at-risk infants early on and ultimately improve survival making use of an early targeted intervention.

ELIGIBILITY:
Inclusion Criteria: Preterm infants with

* Gestational age <28 0/7 weeks
* Birth weight <1000 grams

Exclusion Criteria:

* Major congenital malformations
* Structural airway or lung disease
* Congenital heart disease
* Lack of parental consent

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Presence of pulmonary hypertension | 3-10 days of life (time depending on the timing of the first echocardiography)
  Pulmonary hypertension will be defined as one or more of the following echocardiographic findings:
  * Presence of a cardiac shunt with bidirectional or right-to-left flow
  * Estimated right ventricular systolic pressure (RVSP) >40 mmHg
  * RVSP/systemic systolic blood pressure (SBP) ratio >0.5
  * Presence of ventricular septal wall flattening
Presence of pulmonary hypertension | at 28 days of life
  Pulmonary hypertension will be defined as one or more of the following echocardiographic findings:
  * Presence of a cardiac shunt with bidirectional or right-to-left flow
  * Estimated right ventricular systolic pressure (RVSP) >40 mmHg
  * RVSP/systemic systolic blood pressure (SBP) ratio >0.5
  * Presence of ventricular septal wall flattening
Presence of pulmonary hypertension | at 36 weeks PMA
  Pulmonary hypertension will be defined as one or more of the following echocardiographic findings:
  * Presence of a cardiac shunt with bidirectional or right-to-left flow
  * Estimated right ventricular systolic pressure (RVSP) >40 mmHg
  * RVSP/systemic systolic blood pressure (SBP) ratio >0.5
  * Presence of ventricular septal wall flattening
Presence of pulmonary hypertension | at 6 months of age
  Pulmonary hypertension will be defined as one or more of the following echocardiographic findings:
  * Presence of a cardiac shunt with bidirectional or right-to-left flow
  * Estimated right ventricular systolic pressure (RVSP) >40 mmHg
  * RVSP/systemic systolic blood pressure (SBP) ratio >0.5
  * Presence of ventricular septal wall flattening
Presence of pulmonary hypertension | at 12 months of age
  Pulmonary hypertension will be defined as one or more of the following echocardiographic findings:
  * Presence of a cardiac shunt with bidirectional or right-to-left flow
  * Estimated right ventricular systolic pressure (RVSP) >40 mmHg
  * RVSP/systemic systolic blood pressure (SBP) ratio >0.5
  * Presence of ventricular septal wall flattening

SECONDARY OUTCOMES:
Presence of bronchopulmonary dysplasia | at 28 days of life
  Assessment of supplemental oxygen
Presence of bronchopulmonary dysplasia | at 36 weeks PMA
  Classification of BPD with an oxygen reduction test
Birth weight | at birth
  Birth weight in grams
Gestational age | at birth
  Gestational age in weeks
Small for gestational age | at birth
  Birth weight <P3
Oligohydramnios | at birth
  Presence of oligohydramnios during pregnancy
Maternal hypertensive disorders | at birth
  Presence of maternal hypertensive disorders during pregnancy (pre-eclampsia, hypertension, HELLP)
ROP | at 36 weeks
  Presence of retinopathy of prematurity
NEC | at 36 weeks
  Presence of necrotizing enterocolitis
PDA | at 36 weeks
  Presence of patent ductus arteriosus
Sepsis | up to discharge from the NICU, an average of 16 weeks
  Presence of sepsis
VAP | at 36 weeks
  Presence of ventilator associated pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Barbara De Bisschop, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Filip Cools, PhD, Study Chair — Universitair Ziekenhuis Brussel; Daniël De Wolf, PhD, Study Chair — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arjaans S, Zwart EAH, Ploegstra MJ, Bos AF, Kooi EMW, Hillege HL, Berger RMF. Identification of gaps in the current knowledge on pulmonary hypertension in extremely preterm infants: A systematic review and meta-analysis. Paediatr Perinat Epidemiol. 2018 May;32(3):258-267. doi: 10.1111/ppe.12444. Epub 2018 Jan 17. PMID 29341209
- [Background] Abman SH, Hansmann G, Archer SL, Ivy DD, Adatia I, Chung WK, Hanna BD, Rosenzweig EB, Raj JU, Cornfield D, Stenmark KR, Steinhorn R, Thebaud B, Fineman JR, Kuehne T, Feinstein JA, Friedberg MK, Earing M, Barst RJ, Keller RL, Kinsella JP, Mullen M, Deterding R, Kulik T, Mallory G, Humpl T, Wessel DL; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Surgery and Anesthesia; and the American Thoracic Society. Pediatric Pulmonary Hypertension: Guidelines From the American Heart Association and American Thoracic Society. Circulation. 2015 Nov 24;132(21):2037-99. doi: 10.1161/CIR.0000000000000329. Epub 2015 Nov 3. PMID 26534956
- [Background] Hilgendorff A, Apitz C, Bonnet D, Hansmann G. Pulmonary hypertension associated with acute or chronic lung diseases in the preterm and term neonate and infant. The European Paediatric Pulmonary Vascular Disease Network, endorsed by ISHLT and DGPK. Heart. 2016 May;102 Suppl 2:ii49-56. doi: 10.1136/heartjnl-2015-308591. PMID 27053698
- [Background] Krishnan U, Feinstein JA, Adatia I, Austin ED, Mullen MP, Hopper RK, Hanna B, Romer L, Keller RL, Fineman J, Steinhorn R, Kinsella JP, Ivy DD, Rosenzweig EB, Raj U, Humpl T, Abman SH; Pediatric Pulmonary Hypertension Network (PPHNet). Evaluation and Management of Pulmonary Hypertension in Children with Bronchopulmonary Dysplasia. J Pediatr. 2017 Sep;188:24-34.e1. doi: 10.1016/j.jpeds.2017.05.029. Epub 2017 Jun 20. No abstract available. PMID 28645441
- [Background] Levy PT, Jain A, Nawaytou H, Teitel D, Keller R, Fineman J, Steinhorn R, Abman SH, McNamara PJ; Pediatric Pulmonary Hypertension Network (PPHNet). Risk Assessment and Monitoring of Chronic Pulmonary Hypertension in Premature Infants. J Pediatr. 2020 Feb;217:199-209.e4. doi: 10.1016/j.jpeds.2019.10.034. Epub 2019 Nov 14. No abstract available. PMID 31735418